CLINICAL TRIAL: NCT04419831
Title: Characterizing Subjective and Physiological Responses to Stress and Pain and Cognitive
Brief Title: Characterizing Subjective and Physiological Responses to Stress and Pain and Cognitive Learning and Executive Function
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 2000026626; 000 (Other: CTGTY)
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Pain Response, Stress, Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stress hormones Cortisol and ACTH
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Healthy volunteers: community volunteers
  Interventions: Diagnostic Test: Yale Stress Pain Test (YSPT)
- Binge Heavy drinkers: Individuals who report regular binge alcohol intake and hazardous drinking levels
  Interventions: Diagnostic Test: Yale Stress Pain Test (YSPT)
- Cannabis Use Disorder: Individuals with cannabis use disorder
  Interventions: Diagnostic Test: Yale Stress Pain Test (YSPT)
- Alcohol Use Disorder: Individuals with alcohol use disorder
  Interventions: Diagnostic Test: Yale Stress Pain Test (YSPT)
- Individuals with Moderate to Severe Pain: Individuals with chronic pain
  Interventions: Diagnostic Test: Yale Stress Pain Test (YSPT)
- Opioid Use Disorder in medication assisted treatment: Individuals with opioid use disorder
  Interventions: Diagnostic Test: Yale Stress Pain Test (YSPT)

INTERVENTIONS:
Diagnostic Test: Yale Stress Pain Test (YSPT) — Yale Stress Pain Test involves 10 minutes exposure to 3 cycles of ice cold bucket hand immersion (stress) or 3 cycles of warm water immersion

SUMMARY:
The study design is to assess the between groups factor (controls, chronic pain, addicted individuals) and repeated measures factor of pain/stress (pain vs no pain) along with a longitudinal component to assess stress, pain and addictive behaviors in daily life.

DETAILED DESCRIPTION:
This proposal aims to systematically examine the physiologic, neuroendocrine and behavioral stress and pain responses to an adapted Cold Pressor Test and also assess specific cognitive and executive function tests in community volunteers with a history of stress and trauma, social users of alcohol, cannabis and individuals with alcohol use disorder, cannabis use disorder, opioid use disorder, cocaine use disorder and chronic pain.

ELIGIBILITY:
Inclusion Criteria:

1. Between ages 18-50 years;
2. Able to read and write English;
3. 50 individuals meeting DSM V criteria for Binge Heavy drinkers, using NIAAA criteria for alcohol intake 50 individuals meeting DSM V criteria for Cannabis Use Disorder 50 individuals meeting DSM V criteria for Alcohol Use Disorder 50 Individuals with Moderate to Severe Pain 50 individuals meeting DSM V criteria for Opioid Use Disorder who are initiating treatment
4. Physically healthy as determined by Physical Exam, EKG and blood analyses
5. Body Mass Index (BMI) in the 18-30 range;

Exclusion Criteria:

1. Any psychotic disorder or current psychiatric symptoms requiring specific attention, including active symptoms of psychosis or suicidal/homicidal ideation.
2. Any Current Substance Use Disorder including alcohol, cannabis, cocaine, opioids, sedatives/hypnotics. For alcohol, cannabis, and opioid subjects, exclusion for the abused drug will not apply.
3. Individuals taking any prescription medications or over-the counter medications regularly;
4. Women with irregular menstrual cycles or who are nursing, dysmennorheic, amenorrheic, menopausal, or had premenstrual dysphoric disorder or those on birth control pills;
5. Women who are pregnant as determined by the urine pregnancy test at each laboratory admission;
6. Inability to give informed consent;
7. Traumatic brain injury or loss of consciousness;
8. Individuals with current or past history of seizure disorders

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers and those with chronic pain, those with alcohol use disorder, and those with cannabis use disorder.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Pain assessments | 3 years
  Pain will be assessed by asking participants, "Right now, how much pain do you feel?" asked using the VAS scale ranging from 0 to 100 as outlined in the Laboratory Pain Ratings assessment
Drug craving | 3 years
  Drug craving will be assessed by asking participants, "Right now, how much do you want to use your preferred drug?" This item will be presented in all assessments throughout the study period. Participants will be asked, "How much drug did you use in drinks/grams," that day in the evening prompt and in the previous day in the evening prompt.
Mood and anxiety assessments | 3 years
  The Positive and Negative Affect Schedule (PANAS) measures positive and negative mood and anxiety measures during the initial 28-day period. Participants respond to a 20-item test using a 5-point scale ranging from very slightly or not at all (1) to extremely (5) on the EMA.
Food consumption | 3 years
  Food consumption will be assessed via the evening survey during the initial 28-day period. Participants will respond with the top three types of food that they ate (e.g., "vegetables/salad", "sweet food/dessert", "white meat (e.g., fish/chicken)") and to what extent did they continue eating after feeling full (1=Not at all, 100=Very much).

CONTACTS AND LOCATIONS:
Locations (1):
- Yale Stress Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No